CLINICAL TRIAL: NCT06966232
Title: An Open, Multicentre, Phase 3, Randomized Controlled Clinical Trial to Compare the Prophylactic Use or Preemptive Use of an Anti-viral Drug Entecavir in Patients With Gastrointestinal Cancer Who Are Inactive Hepatitis B Carriers
Brief Title: Prophylactic or Preemptive Entecavir in Patients With Gastrointestinal Cancer Who Are Inactive Hepatitis B Carriers
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Rui-hua Xu, MD, PhD, The president of Sun Yat-sen University Cancer Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIC-HBV
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Gastrointestinal Cancers
Keywords: Gastrointestinal Cancers; Entecavir; Hepatitis B Carrier; Chemotherapy; Immunotherapy
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic Entecavir (Experimental): Entecavir is prophylactically used from the time of chemotherapy or immunotherapy initiation at the dose of 0.5 mg p.o daily till 6 months after the end of chemotherapy or immunotherapy .
  Interventions: Drug: Entecavir
- Preemptive Entecavir (Active Comparator): Entecavir is preemptively used from the time that hepatitis B virus DNA copies become positive at the dose of 0.5 mg p.o daily till 6 months after the end of chemotherapy or immunotherapy.
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Entecavir — anti hepatitis B virus
  Other Names: Entecavir Dispersible Tablets

SUMMARY:
There has been no report on whether the patients with gastrointestinal cancer who are also inactive hepatitis B carriers should receive prophylactic use or preemptive use of an anti-viral drug entecavir during anti-tumor therapy. This open, multicentre, phase 3, randomized controlled clinical trial aims to compare the impact of the prophylactic use or preemptive use of an anti-viral drug entecavir on the outcomes of patients with gastrointestinal cancer who are also inactive hepatitis B carriers during chemotherapy or immunotherapy and the subsequent follow-ups, including two cohorts of chemotherapy and immunotherapy.

DETAILED DESCRIPTION:
Patients with gastrointestinal cancer who are also inactive hepatitis B carriers are enrolled and randomized into two groups as following. Patients in experimental group are treated with entecavir prophylactically in the dose of 0.5mg p.o. every day from the initiation of chemotherapy or immunotherapy till 6 months after the end of chemotherapy or immunotherapy. Patients in active comparator group are only treated with entecavir in the dose of 0.5mg p.o. every day from the time that the DNA copies of hepatitis B virus become positive till 6 months after the end of chemotherapy or immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with age between 18 and 75
2. Patient with histology-proven locally advanced unresectable or metastatic gastrointestinal cancers (colorectal cancer, gastric cancer, esophageal cancer, hepatocellular carcinoma, pancreatic cancer, and cholangiocarcinoma)
3. Planned to receive first-, second-, or third-line anti-tumor therapy (chemotherapy or PD-1/PD-L1 monoclonal antibody immunotherapy)
4. Patients with Eastern Cooperative Oncology Group performance status (ECOG) of 0-2
5. Patients planned for at least 4 cycles of chemotherapy or immunotherapy
6. Patients with at least 6 months' life expectancy from date of recruitment
7. Patients with chronic or past HBV infection (HBsAg-positive or HBcAb-positive), and hepatitis B is inactive
8. Patients with normal liver function tests including alanine aminotransferase (ALT), aspartate aminotransferase alkaline (AST), and bilirubin
9. Patients with negative HBV-DNA
10. Adequate major organ function (laboratory tests 14 days before randomization meeting requirements for anti-tumor therapy)
11. Patients who sign the informed consent
12. Patients with good compliance during chemotherapy and follow-ups.

Exclusion Criteria:

1. History of liver cirrhosis
2. Prior HBV reactivation
3. Received anti-HBV therapy for chronic hepatitis B within 6 months before enrollment
4. Active co-infection with other hepatitis viruses
5. HIV infection
6. Autoimmune hepatitis
7. History of hepatic radiotherapy
8. Scheduled hepatic radiotherapy or radioisotope therapy
9. Pregnant or lactating women
10. Patients with a history of psychiatric drugs abuse and can't quit or with a mental disorder
11. Patients with immunodeficiency, other congenital or acquired immunodeficiency, or transplantation history
12. According to the investigators' judgment, patients with concomitant disease that seriously harms patients' safety or the completion of study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-05-20 (Estimated)

PRIMARY OUTCOMES:
The incidence of hepatitis B virus reactivation | through study completion, an average of 1 year
  HBV reactivation is defined as (1) an increase in HBV-DNA levels by ≥2 log10 (100-fold) compared to baseline or conversion from negative serum HBV-DNA to positive HBV-DNA; (2) if baseline HBV-DNA was undetectable, achieving HBV-DNA levels ≥3 log10 (1,000 IU/mL); or (3) if baseline levels were unknown or unavailable, reaching HBV-DNA levels ≥4 log10 (10,000 IU/mL).

SECONDARY OUTCOMES:
Hepatitis | through study completion, an average of 1 year
  Hepatitis is defined as a 3-fold or greater increase in the serum ALT level that exceeded the reference range or an absolute increase in the level of ALT of greater than 100 U/L compared with the baseline level
Hepatitis B virus associated hepatitis | through study completion, an average of 1 year
  Hepatitis B virus associated hepatitis is defined as hepatitis B virus (HBV) reactivation occurring prior to or concurrent with hepatitis during or following chemotherapy/immunotherapy , in the absence of clinical or laboratory evidence of acute infection by other hepatitis viruses or systemic diseases.
Interruption of chemotherapy/immunotherapy due to hepatitis | through study completion, an average of 1 year
  Chemotherapy/immunotherapy disruption due to hepatitis is defined as either premature termination or a delay of at least 7 days between therapy cycles due to hepatitis .
Severe HBV associated hepatitis | through study completion, an average of 1 year
  Severe HBV associated hepatitis is defined as grade 3 or higher HBV associated hepatitis according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
HBV associated acute liver failure | through study completion, an average of 1 year
  HBV associated acute liver failure, also termed HBV associated fulminant hepatic failure , is defined as acute hepatic decompensation linked to HBV reactivation or acute exacerbation of HBV infection. It manifests within days to weeks, leading to severe complications such as coagulopathy, hepatic encephalopathy, and multiorgan failure, with a high 28-day mortality rate . Delayed initiation of nucleotide analogues may contribute to rapid disease progression and poor prognosis.
HBV related death | through study completion, an average of 1 year
  HBV related death is defined as mortality directly attributable to HBV reactivation

CONTACTS AND LOCATIONS:
Overall Officials: Xu Rui-hua, M.D. Ph.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Perrillo RP, Gish R, Falck-Ytter YT. American Gastroenterological Association Institute technical review on prevention and treatment of hepatitis B virus reactivation during immunosuppressive drug therapy. Gastroenterology. 2015 Jan;148(1):221-244.e3. doi: 10.1053/j.gastro.2014.10.038. Epub 2014 Oct 31. No abstract available. PMID 25447852
- [Background] Huang H, Li X, Zhu J, Ye S, Zhang H, Wang W, Wu X, Peng J, Xu B, Lin Y, Cao Y, Li H, Lin S, Liu Q, Lin T. Entecavir vs lamivudine for prevention of hepatitis B virus reactivation among patients with untreated diffuse large B-cell lymphoma receiving R-CHOP chemotherapy: a randomized clinical trial. JAMA. 2014 Dec 17;312(23):2521-30. doi: 10.1001/jama.2014.15704. PMID 25514302